CLINICAL TRIAL: NCT03436017
Title: Identification of Biomarkers of Attention Deficit Disorder With or Without Hyperactivity (ADHD) by a Metabolomic Approach in Children
Acronym: METHADA
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI17/METHADA
Record Dates: First submitted 2018-01-24; First posted 2018-02-19 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Adhd
Keywords: adhd; metabolomics; child
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples Urinary samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD: Patient with ADHD diagnosis criterion. The aim is the identification of Biomarkers of ADHD by a Metabolomic Approach
  Interventions: Other: Metabolomic approach
- non ADHD: Patient with symptom of hyperactivity and/or attention deficiency but without ADHD diagnosis criterion.
  The aim is the identification of Biomarkers of ADHD by a Metabolomic Approach.
  Interventions: Other: Metabolomic approach

INTERVENTIONS:
Other: Metabolomic approach — Biological samples (blood and urine) for a multimodal metabolomic approach

SUMMARY:
Attention-deficit with or without hyperactivity disorder (ADHD) is a real health public concern. No easy-use diagnosis tool are available. Metabolomic approaches has brought very usefull data in others neurological diseases like amyotrophic lateral sclerosis or autism spectrum disorder, as we had shown in previous studies. Targeting on neurotransmitter pathways involving in ADHD, metabolomic screening could help to enhance our diagnosis power to better help numerus of children. We propose to study the phenylalanine and the tyrosine pathways with a multimodal metabolomic approach, in easy-available biological fluid (blood and urine), in child or adolescent suspected of ADHD. Our objectives are: 1- to determine a specific metabolomic signature of ADHD 2- to compare the diagnostic value of this metabolomic signature with the reference methodology for ADHD diagnosis, as now practiced in our reference center for learning troubles.

ELIGIBILITY:
Inclusion Criteria:

* Child or adolescent with symptoms of attention disorders and / or hyperactivity
* aged from 6 to 15 years old

Exclusion Criteria:

* Failure or refusal of all or part of the multidisciplinary evaluation (medical and / or neuropsychological assessments and / or biological assessments)
* Identification of an intercurrent condition likely to have an impact on metabolomic analyzes (acute infection, fever, etc.)
* Parents or legal guardians opposed to data processing

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child or adolescent with symptoms of attention disorders and / or hyperactivity, aged from 6 to 15 years old, and consulting in current care in our university hospital
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
ADHD metabolomic's signature of blood | At baseline
  Detection of metabolites (phenylalanine or catécholamines) in the blood of patients with ADHD at levels significantly different from baseline levels in the general population and rates found in patients with attention deficit and / or hyperactivity disorders but that multidisciplinary assessment excludes the diagnosis of ADHD.
ADHD metabolomic's signature of urine | At baseline
  Detection of metabolites (phenylalanine or catécholamines) in the urine of patients with ADHD at levels significantly different from baseline levels in the general population and rates found in patients with attention deficit and / or hyperactivity disorders but that multidisciplinary assessment excludes the diagnosis of ADHD.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CASTELNAU, MD-PhD, Principal Investigator — CHU Tours
Locations (1):
- University Hospital TOURS, Tours, France